CLINICAL TRIAL: NCT01221727
Title: The Effects of Denosumab on the Pharmacokinetics (PK) of Midazolam, a Cytochrome P450 3A4/P-gp (CYP3A4) Substrate, in Postmenopausal Osteoporotic Women
Brief Title: The Effects of Denosumab on the Pharmacokinetics (PK) of Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20101131
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2015-09

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Amgen; Phase 1; Postmenopausal; Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Denosumab; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam (Other): All 27 subjects will receive midazolam.
  Interventions: Drug: Denosumab
- Denosumab (Active Comparator): Eighteen (18) subjects will receive denosumab.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Denosumab — Eighteen (18) subjects will receive 1 fixed dose administration of denosumab.
  Other Names: AMG 162
  Arms: Midazolam
Drug: Midazolam — All subjects will receive two oral dose administrations of midazolam.
  Arms: Denosumab

SUMMARY:
This is a multi-center, open-label, drug-drug interaction study in postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
Approximately 27 subjects (Group A: 18; Group B: 9) will receive a 2 mg oral dose of midazolam on day 1 followed by a 24 hour PK collection. Subjects randomized to Group A will receive a single 60 mg subcutaneous (SC) dose of denosumab on day 2 administered in the abdomen. On study day 16, another 2 mg oral dose of midazolam will be administered to all subjects (Groups A and B) followed by a 24 hour PK collection. The primary analysis to determine the effect of denosumab on the PK of midazolam will be based on data from subjects in Group A only.

ELIGIBILITY:
Inclusion Criteria:

* Between 45 to 75 years of age
* Postmenopausal women
* Osteoporosis

Exclusion Criteria:

* Use of any known inhibitors of cytochrome P450 3A4/P-gp (CYP3A4) within 14 days or 5 half lives, whichever is longer; or grapefruit juice or grapefruit containing products within 7 days prior to investigational product administration
* Use of any known CYP3A4 inducers within 30 days or 5 half-lives, whichever is longer, prior to investigational product administration
* Use of any herbal medicine with a known impact on CYP3A4 (eg, St. John's wort) within 30 days prior to investigational product administration
* Current use of medications prescribed for osteoporosis treatment
* Use of midazolam within 14 days prior to investigational product administration
* Influenza or other vaccination within 28 days of screening
* Previous exposure to denosumab

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Jang G, Kaufman A, Lee E, Hamilton L, Hutton S, Egbuna O, Padhi D. A clinical therapeutic protein drug-drug interaction study: coadministration of denosumab and midazolam in postmenopausal women with osteoporosis. Pharmacol Res Perspect. 2014 Apr;2(2):e00033. doi: 10.1002/prp2.33. Epub 2014 Mar 13. PMID 25505582
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Midazolam With Denosumab: 2 mg oral dose of Midazolam on Day 1 and Day 16, 60 mg subcutaneous dose of Denosumab on Day 2
- Midazolam Only: 2 mg oral dose of Midazolam on Day 1 and Day 16.
Period: Overall Study
Arm/Group | Midazolam With Denosumab | Midazolam Only
Started | 21 (Number of subjects randomized into the study) | 9 (Number of subjects randomized into the study)
Treated | 19 (Number of subjects received investigational product) | 8 (Number of subjects received investigational product)
Completed | 18 | 8
Not Completed | 3 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Midazolam With Denosumab: 2 mg oral dose of Midazolam on Day 1 and Day 16, 60 mg subcutaneous dose of Denosumab on Day 2. Out of 21 subjects enrolled and randomized, 19 subjects received investigation product.
- Midazolam Only: 2 mg oral dose of Midazolam on Day 1 and Day 16. Out of 9 subjects enrolled and randomized, 8 subjects received investigation product.
- Total: Total of all reporting groups
Arm/Group | Midazolam With Denosumab | Midazolam Only | Total
Number analyzed (Participants) | 19 | 8 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.42 (6.16) | 66.25 (5.34) | 64.96 (5.89)
Age, Customized [Number; unit: Participants]
  <65 years | 7 | 3 | 10
  >=65 years and <75 years | 12 | 4 | 16
  >=75 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 8 | 27
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 12 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 6 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Pharmcokinetic (PK) Area Under the Concentration Time Curve (AUC) Parameter Estimates Between Day 16 (Midazolam With the Presence of Denosumab) and Day 1 (Midazolam Only)
Description: The ratio and confidence interval are calculated based on natural log scale data and converted back to the original scale.
Time Frame: From day 1 pre-dose to 24 hours post-dose and from day 16 pre-dose to 24 hours post-dose
Population: The analysis set will contain all subjects from Midazolam with Denosumab group for whom the primary endpoint PK parameters (AUC(0-t), AUC(0-inf) and Cmax) can be estimated for both treatment periods.
Measure: Least Squares Mean (90% Confidence Interval); unit: unitless
Units Other Than Participants: unitless
Groups:
- Midazolam With Denosumab: Subjects received 2 mg oral dose of Midazolam on day 1 (serving as a reference point) and day 16 (serving as a test point), and 60 mg subcutaneous dose of Denosumab on day 2
Arm/Group | Midazolam With Denosumab
Number analyzed (Participants) | 18
Number analyzed (unitless) | 18
unitless
  AUC (0-t) | 1.10 [0.94 to 1.29]
  AUC (0-inf) | 1.12 [0.95 to 1.31]

2. Secondary Outcome: Ratio of PK AUC Parameter Estimates Between Day 16 (Midazolam Only) and Day 1(Midazolam Only)
Description: as for outcome 1
Time Frame: From day 1 pre-dose to 24 hours post-dose and from day 16 pre-dose to 24 hours post-dose
Population: The analysis set will contain all subjects from Midazolam only group for whom the primary endpoint PK parameters (AUC(0-t), AUC(0-inf) and Cmax) can be estimated for both treatment periods.
Measure: Least Squares Mean (90% Confidence Interval); unit: unitless
Units Other Than Participants: unitless
Groups:
- Midazolam Only: Subjects received 2 mg oral dose of Midazolam on day 1 and day 16
Arm/Group | Midazolam Only
Number analyzed (Participants) | 8
Number analyzed (unitless) | 8
unitless
  AUC (0-t) | 0.98 [0.83 to 1.15]
  AUC (0-inf) | 0.98 [0.84 to 1.15]

3. Primary Outcome: Estimates of Inter- and Intra-subject Variability for the PK AUC Parameters for Midazolam With Denosumab Group
Description: AUC Subject denotes the inter-subject variability, while AUC Residual denotes the intra-subject variability
Time Frame: From day 1 pre-dose to 24 hours post-dose and from day 16 pre-dose to 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Units Other Than Participants: area
Groups:
- Midazolam With Denosumab: Subjects received 2 mg oral dose of Midazolam on day 1 and day 16 , and 60 mg subcutaneous dose of Denosumab on day 2
Arm/Group | Midazolam With Denosumab
Number analyzed (Participants) | 18
Number analyzed (area) | 18
ng*hr/mL
  AUC (0-t) Subject: Inter-subject | 0.19 (0.079)
  AUC (0-t) Residual: Intra-subject | 0.07 (0.025)
  AUC (0-inf) Subject: Inter-subject | 0.21 (0.085)
  AUC (0-inf) Residual: Intra-subject | 0.08 (0.027)

4. Primary Outcome: Estimates of Inter- and Intra-subject Variability for PK Maximum Observed Plasma Concentration (Cmax) Parameter for Midazolam With Denosumab Group
Description: Cmax Subject denotes the inter-subject variability, while Cmax Residual denotes the intra-subject variability
Time Frame: From day 1 pre-dose to 24 hours post-dose and from day 16 pre-dose to 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: concentration
Groups:
- Midazolam With Denosumab: Subjects received 2 mg oral dose of Midazolam on day 1 and day 16, and 60 mg subcutaneous dose of Denosumab on day 2
Arm/Group | Midazolam With Denosumab
Number analyzed (Participants) | 18
Number analyzed (concentration) | 18
ng/mL
  Cmax Subject: Inter-subject | 0.15 (0.064)
  Cmax Residual: Intra-subject | 0.07 (0.023)

5. Secondary Outcome: Estimates of Inter- and Intra-subject Variability for the PK AUC Parameters for Midazolam Only Group
Description: AUC Subject denotes the inter-subject variability, while AUC Residual denotes the intra-subject variability.
Time Frame: From day 1 pre-dose to 24 hours post-dose and from day 16 pre-dose to 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Units Other Than Participants: area
Arm/Group | Midazolam Only
Number analyzed (Participants) | 8
Number analyzed (area) | 8
ng*hr/mL
  AUC (0-t) Subject: Inter-subject | 0.27 (0.155)
  AUC (0-t) Residual: Intra-subject | 0.03 (0.016)
  AUC (0-inf) Subject: Inter-subject | 0.31 (0.175)
  AUC (0-inf) Residual: Intra-subject | 0.03 (0.015)

6. Secondary Outcome: Estimates of Inter- and Intra-subject Variability for PK Cmax Parameter for Midazolam Only Group
Description: Cmax Subject denotes the inter-subject variability, while Cmax Residual denotes the intra-subject variability.
Time Frame: From day 1 pre-dose to 24 hours post-dose and from day 16 pre-dose to 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: concentration
Arm/Group | Midazolam Only
Number analyzed (Participants) | 8
Number analyzed (concentration) | 8
ng/mL
  Cmax Subject: Inter-subject | 0.23 (0.143)
  Cmax Residual: Intra-subject | 0.06 (0.035)

7. Secondary Outcome: Summary of Serum Denosumab Concentration
Description: This table summarizes serum Denosumab for Midazolam with Denosumab group. The Lower Limit Of Quantification (LLOQ) is 20 ng/mL. On Day 2 (pre-dose), the true value is below LLOQ, and is treated as 0 in the analysis.
Time Frame: Baseline (day 2 pre-dose) to day 16
Population: Serum Denosumab will be collected for subjects in Midazolam with Denosumab group only. The analysis set will contain subjects in Midazolam with Denosumab group who received denosumab administration and for whom serum Denosumab concentrations are determinable when assessed.
Measure: Median (Standard Deviation); unit: ng/mL
Units Other Than Participants: concentration
Arm/Group | Midazolam With Denosumab
Number analyzed (Participants) | 18
Number analyzed (concentration) | 18
ng/mL
  Day 2 (Pre-dose) | 0 (NA) — All the pre-dose concentration measurements are below LLOQ, and were treated as 0 in the analysis. Therefore, the true standard deviation is not able to be calculated.
  Day 16 (0hr) | 5820 (1800)
  Day 17 (24hr) | 5500 (1940)

8. Secondary Outcome: Summary of Serum C-Telopeptide Concentration
Description: This table summarizes serum C-Telopeptide (sCTX) concentration raw values for Midazolam with Denosumab group.
Time Frame: Baseline (day 2 pre-dose) to day 16
Population: Serum CTX will be collected for Midazolam with Denosumab group only. The PD analysis set will contain subjects in Midazolam with Denosumab group who received denosumab administration and for whom serum CTX concentrations are determinable on when assessed.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Units Other Than Participants: concentration
Arm/Group | Midazolam With Denosumab
Number analyzed (Participants) | 18
Number analyzed (concentration) | 18
ng/mL
  Baseline (day 2 pre-dose) | 0.4655 (0.0698) [0.3390 to 0.6290]
  Day 16 | 0.0606 (0.0030) [0.0483 to 0.0662]
  Change from baseline to Day 16 | -0.4079 (0.0702) [-0.5752 to -0.2712]

9. Primary Outcome: Ratio of PK Cmax Parameter Estimates Between Day 16 (Midazolam With the Presence of Denosumab) and Day 1 (Midazolam Only)
Description: as for outcome 1
Time Frame: From day 1 pre-dose to 24 hours post-dose and from day 16 pre-dose to 24 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: unitless
Units Other Than Participants: unitless
Arm/Group | Midazolam With Denosumab
Number analyzed (Participants) | 18
Number analyzed (unitless) | 18
unitless | 1.11 [0.96 to 1.29]

10. Secondary Outcome: Summary of Percent Change From Baseline to Day 16 for Serum C-Telopeptide Concentration
Description: This table summarizes percent change from baseline to day 16 for serum C-Telopeptide (sCTX) concentration raw values for Midazolam with Denosumab group.
Time Frame: Baseline (day 2 pre-dose) to day 16
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: percentage
Units Other Than Participants: percentage
Arm/Group | Midazolam With Denosumab
Number analyzed (Participants) | 18
Number analyzed (percentage) | 18
percentage | -87.52 [-91.45 to -80.01]

11. Secondary Outcome: Ratio of PK Cmax Parameter Estimates Between Day 16 (Midazolam Only) and Day 1(Midazolam Only)
Description: as for outcome 1
Time Frame: From day 1 pre-dose to 24 hours post-dose and from day 16 pre-dose to 24 hours post-dose
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: unitless
Units Other Than Participants: unitless
Arm/Group | Midazolam Only
Number analyzed (Participants) | 8
Number analyzed (unitless) | 8
unitless | 1.05 [0.82 to 1.33]

ADVERSE EVENTS:
Time Frame: 47 days
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Midazolam With Denosumab Group With Midazolam 2mg on Day 1 | Midazolam With Denosumab Group With Denosumab 60mg on Day 2-15 | Midazolam With Denosumab Group With Midazolam 2mg on Day 16 | Midazolam Only Group With Midazolam 2mg on Day 1 | Midazolam Only Group With Midazolam 2mg on Day 2-15 | Midazolam Only Group With Midazolam 2mg on Day 16
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/18 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 9/19 | 6/18 | 10/18 | 2/8 | 1/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Midazolam With Denosumab Group With Midazolam 2mg on Day 1 (N=19) | Midazolam With Denosumab Group With Denosumab 60mg on Day 2-15 (N=18) | Midazolam With Denosumab Group With Midazolam 2mg on Day 16 (N=18) | Midazolam Only Group With Midazolam 2mg on Day 1 (N=8) | Midazolam Only Group With Midazolam 2mg on Day 2-15 (N=8) | Midazolam Only Group With Midazolam 2mg on Day 16 (N=8)
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 3 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 7 | 0 | 7 | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.